CLINICAL TRIAL: NCT00085449
Title: A Trial of Reduced Intensity Conditioning and Transplantation of Haplotype Mismatched and KIR Class I Epitope-Mismatched Highly Purified CD34 Cells
Brief Title: Alemtuzumab Plus Fludarabine and Melphalan With or Without Cyclosporine, Mycophenolate Mofetil, and Low-Dose Total-Body Irradiation Therapy Followed by Donor Peripheral Stem Cell Transplant in Treating Patients With Hematologic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding cut, no patients enrolled
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-100102; CALGB-100102; CDR0000370797 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission; recurrent adult acute lymphoblastic leukemia; adult acute lymphoblastic leukemia in remission; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; chronic myelomonocytic leukemia; recurrent adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent small lymphocytic lymphoma; recurrent marginal zone lymphoma; recurrent mantle cell lymphoma; recurrent adult lymphoblastic lymphoma; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory multiple myeloma; secondary myelodysplastic syndromes; de novo myelodysplastic syndromes; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Lymphoma, Large B-Cell, Diffuse; Congenital Abnormalities | interventions — Alemtuzumab; Cyclosporine; fludarabine phosphate; Melphalan; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regimen A + B (Experimental): Conditioning regimen A: Patients receive alemtuzumab IV over 2 hours on days -14 to -12; fludarabine IV over 30 minutes on days -7 to -3; and melphalan IV over 20-30 minutes on day -2.
  Conditioning regimen B: Patients receive oral or IV cyclosporine twice daily and oral or IV mycophenolate mofetil twice daily on days -15 to 0. Patients also receive alemtuzumab, fludarabine, and melphalan as in conditioning regimen A. Patients undergo low-dose total body irradiation twice daily on days -2 and -1.
  All patients undergo allogeneic, T-cell-depleted, CD34-positive peripheral blood stem cell transplantation on day 0. Patients receive sargramostim (GM-CSF) subcutaneously beginning on day 1 and continuing until blood counts recover.
  Patients are followed every 3 months for 1 year and then every 6 months for 5 years.
  Interventions: Biological: alemtuzumab; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: melphalan; Drug: mycophenolate mofetil; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: alemtuzumab
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: melphalan
Drug: mycophenolate mofetil
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, monoclonal antibodies, and radiation therapy before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells when they do not exactly match the patient's blood. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil before transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects of alemtuzumab, fludarabine, and melphalan with or without cyclosporine, mycophenolate mofetil, and total-body irradiation before donor peripheral blood stem cell transplant and to see how well they work in treating patients with relapsed or refractory hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability of a reduced-intensity conditioning regimen comprising alemtuzumab, fludarabine, and melphalan with or without cyclosporine, mycophenolate mofetil, and low-dose total body radiotherapy followed by haplotype-mismatched, KIR class I epitope-mismatched CD34-positive allogeneic peripheral blood stem cell transplantation to facilitate engraftment by day 35 post-transplantation in at least 85% of patients with relapsed, refractory, or poor-risk hematological malignancies.
* Determine the risk of graft-versus-host-disease in patients treated with these regimens.
* Determine, preliminarily, the efficacy of these regimens, in terms of progression-free survival, in these patients.
* Correlate outcomes, engraftment, and progression-free survival with the number of detectable alloreactive natural killer cell clones before transplantation and after engraftment in patients treated with these regimens.
* Determine immune reconstitution in patients treated with these regimens.

OUTLINE: This is a multicenter, pilot study. Patients are initially treated with conditioning regimen A. If adequate donor engraftment is not achieved, subsequent patients are treated with conditioning regimen B.

* Conditioning regimen A: Patients receive alemtuzumab IV over 2 hours on days -14 to -12; fludarabine IV over 30 minutes on days -7 to -3; and melphalan IV over 20-30 minutes on day -2.
* Conditioning regimen B: Patients receive oral or IV cyclosporine twice daily and oral or IV mycophenolate mofetil twice daily on days -15 to 0. Patients also receive alemtuzumab, fludarabine, and melphalan as in conditioning regimen A. Patients undergo low-dose total body irradiation twice daily on days -2 and -1.

All patients undergo allogeneic, T-cell-depleted, CD34-positive peripheral blood stem cell transplantation on day 0. Patients receive sargramostim (GM-CSF) subcutaneously beginning on day 1 and continuing until blood counts recover.

Patients are followed every 3 months for 1 year and then every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 14-56 patients (14-28 per regimen) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hematological malignancy of 1 of the following types:

  * Acute myeloid leukemia meeting at least 1 of the following criteria:

    * Poor-risk cytogenetics, including -5, 5q-, -7, 7q-, 11q23, and Philadelphia (Ph) chromosome-positive in first or subsequent complete remission (CR)
    * Relapsed or primary refractory disease with ≤ 10% blasts in the peripheral blood and ≤ 20% blasts in the bone marrow
    * Standard-risk cytogenetics in second CR AND autologous transplantation is not feasible
    * Standard-risk cytogenetics in third or subsequent CR
  * Acute lymphoblastic leukemia meeting 1 of the following criteria:

    * Second or subsequent CR
    * High-risk cytogenetics, including Ph chromosome-positive and t(4:11) in first CR
    * Relapsed or primarily refractory disease with ≤ 10% blasts in the peripheral blood and ≤ 20% blasts in the bone marrow
  * High-risk myelodysplasia

    * International Prognostic Scoring System Score ≥ 2.5
  * Chronic myeloid leukemia (CML)* with an inadequate response to imatinib meeting 1 of the following criteria:

    * Second or subsequent chronic phase
    * Accelerated phase NOTE: *Patients with CML in blast crisis (> 30% promyelocytes and myeloblasts in the bone marrow) are not eligible
  * Non-Hodgkin's lymphoma meeting 1 of the following criteria:

    * Primarily refractory disease or in refractory relapse
    * Relapsed disease after autologous stem cell transplantation
    * Chemosensitive relapsed disease without CR to standard salvage therapy AND no option for autologous stem cell transplantation due to blood or marrow involvement or failure to harvest sufficient autologous stem cells
  * Chronic lymphocytic leukemia meeting both of the following criteria:

    * Stage III or IV disease
    * Refractory to fludarabine
  * Multiple myeloma meeting 1 of the following criteria:

    * Primarily refractory disease or in refractory relapse
    * Relapsed disease after autologous stem cell transplantation
* No relapsed disease < 6 months after autologous stem cell transplantation
* No available eligible HLA-matched (i.e., 5 of 6 or 6 of 6 antigen match for HLA-A, -B, and -DR loci) family donor by serological or molecular typing
* Available suitable family donor meeting the following criteria:

  * Parent, sibling, or child of the recipient
  * ≥ 16 years of age
  * Identical for only one HLA haplotype (i.e., haploidentical) AND incompatible at the HLA-A, -B, -C, and -DR loci of the unshared haplotype by serological or molecular typing
  * Mismatched with respect to KIR class I epitopes graft-vs-host directional activity

    * Mismatching that predicts both graft-vs-host and host-vs-graft bi-directional activity eligible
    * No mismatching that predicts only host-vs-graft directional activity

PATIENT CHARACTERISTICS:

Age

* 18 to 60

Performance status

* ECOG 0-1

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* AST and ALT < 2 times ULN

Renal

* Creatinine ≤ 2 mg/dL

Cardiovascular

* LVEF > 40% (corrected)

Pulmonary

* DLCO > 50% of predicted

Other

* No active infection requiring oral or IV antibiotics
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Concurrent corticosteroids allowed for adrenal failure, treatment of graft-vs-host disease, or as premedication during study
* No concurrent corticosteroids for antiemesis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Engraftment rate | Up to 6 years
Risk of graft-vs-host disease | Up to 6 years
Progression-free survival (PFS) | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Sherif S. Farag, MD, PhD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (24):
- United States (24):
  - Moores UCSD Cancer Center, La Jolla, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia